CLINICAL TRIAL: NCT03153553
Title: Ischemic Preconditioning, Exercise Tolerance and Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STH19739
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischaemic Preconditioning Group (Active Comparator): The participant will rest in a sitting position for 10 minutes before measuring resting blood pressure. Blood pressure will be measured on the arm. IPC will be administered to the upper arm using cuff inflation pressures of 30mm Hg above the systolic BP using a manual BP. The IPC cycles comprised of three cycles of cuff inflation each lasting 5 min in duration followed by 5-min period of cuff deflation
  Interventions: Other: Ischemic Preconditioning
- Control group (Sham Comparator): The participant will rest in a sitting position for 10 min before measuring resting blood pressure. Blood pressure will be measured on the upper arm. Sham intervention will be administered to the right upper limb using a manual BP cuff which will be inflated at a pressure 30mmg Hg below the diastolic blood pressure. The sham cycles comprised of three cycles of cuff inflation each lasting 5 minutes in duration followed by 5-min period of cuff deflation
  Interventions: Other: Sham Intervention

INTERVENTIONS:
Other: Ischemic Preconditioning — Ischemic preconditioning (IPC) is an experimental technique for producing resistance to the loss of blood supply, and thus oxygen, to tissues of many types. In the heart, IPC is an intrinsic process whereby repeated short episodes of ischaemia protect the myocardium against a subsequent ischaemic insult
  Arms: Ischaemic Preconditioning Group
Other: Sham Intervention — Sham intervention will be administered to the right upper limb using a manual BP cuff which will be inflated at a pressure 30mmg Hg below the diastolic blood pressure. The sham cycles comprised of three cycles of cuff inflation each lasting 5 minutes in duration followed by 5-min period of cuff deflation
  Arms: Control group

SUMMARY:
Regular physical activity improves aspects such as physical fitness, fatigue, quality of life, gait and also reduces the rate of progression of disability in individuals with Multiple Sclerosis. However, individuals with multiple sclerosis are less physically active than the general population. The determinants of engaging in physical activity for individuals with multiple sclerosis include psychological factors like motivation, self-belief and self-regulatory constructs and physical factors like fatigue, weakness, pain and ataxia.

Ischemic preconditioning is exposure of the body to brief periods of circulatory occlusion and re-perfusion to protect organs against ischemic injury. Recent studies have also shown that ischemic preconditioning also improves exercise performance in healthy participants.

The primary aim and objective of this study is to see whether it is feasible to use Ischemic preconditioning to improve exercise performance in people with Multiple Sclerosis.

The design for the study is a double blind randomized control trial. Forty patients with multiple sclerosis above 18 years of age and who have the ability to walk will be randomized to receive either Ischemic preconditioning or sham intervention. All participants will be identified by MS consultants and nurses from the MS clinic and Neuro Day Case Unit of the Royal Hallamshire Hospital in Sheffield. Participation will involve an additional 2 hours of the patients time.

DETAILED DESCRIPTION:
This project is quantified as a Feasibility study. The design for the study is a double blind randomised control trial. Forty patients with MS above 18 years and who have the ability to walk will be randomised to receive either IPC or sham intervention. Potential candidates will be identified from the MS clinic and Neuro Day Case Unit of the Royal Hallamshire Hospital (RHH) in Sheffield.

All participants will be identified by MS consultants and nurses from MS clinics and from neuroday case unit of Royal Hallamshire Hospital. The patient information sheet will be mailed to the participants deemed suitable for the trial by the treating team. The participants will be given up to two weeks to consider their participation in the trial. Patients wishing to participate will be consented by Dr Siva Nair/Kate Lavender/Dr Ismail, following consent Dr Nair/Kate Lavender/ Dr Ismail will ensure the participants are randomised into the treatment group or the control group using a random number table. The MSc student will act as blinded assessor.

After obtaining consent, the research team will conduct checks against the inclusion criteria to assess whether the participant fulfils the criteria for entry into the study. The participant will then be allocated into one of the two groups using a random number table: Experimental group or the Sham group. Participants will not be told which group they have been randomised to. The researcher will check the participant's blood pressure and heart rate while sitting. Then the researcher will request the participant to walk for six minutes as they normally walk. The researcher will measure the distance covered in 6 minutes and will ask the participant to grade the exertion experienced using Borg's Rating of Perceived Exertion scale. The researcher will again measure the blood pressure and heart rate again.

In the active comparator group The participant will rest in a sitting position for 10 minutes before measuring resting blood pressure. Blood pressure will be measured on the arm. IPC will be administered to the upper arm using cuff inflation pressures of 30mm Hg above the systolic BP using a manual BP. The IPC cycles comprised of three cycles of cuff inflation each lasting 5 min in duration followed by 5-min period of cuff deflation.

Within the sham intervention The participant will rest in a sitting position for 10 min before measuring resting blood pressure. Blood pressure will be measured on the upper arm. Sham intervention will be administered to the right upper limb using a manual BP cuff which will be inflated at a pressure 30mmg Hg below the diastolic blood pressure. The sham cycles comprised of three cycles of cuff inflation each lasting 5 minutes in duration followed by 5-min period of cuff deflation.

The researcher will ask the participant to grade any pain or discomfort experienced during the intervention in a scale of 0 (no pain or discomfort) to 10 (Worst pain or discomfort ever experience).

Ten minutes after the end of the cycle the Researcher will again measure the blood pressure and heart rate. Then the participant will be asked to walk for six minutes with the researcher. The researcher will measure the distance covered in 6 minutes. The researcher will ask the participant to grade the exertion experienced using Rating of Perceived Exertion. The researcher will measure the blood pressure and heart rate again. We anticipate that the patient spend around 2 hours at Royal Hallamshire Hospital for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MS as per the McDonald's criteria
2. Aged 18 or older
3. Sufficient cognitive ability to give informed consent
4. Ability to walk for 6 minutes without rest
5. Resting Systolic BP of less than 170 mmHg

Exclusion Criteria:

1. Cognitive difficulties in giving consent ad understanding the questionnaire
2. Inability to walk
3. Other systemic illness affecting exercise tolerance
4. Resting systolic BP of 170mmHg or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Ability to tolerate Ischaemic Preconditioning (IPC_ | One day
  Patients will be asked to indicate the tolerability of IPC using a visual analogue scale from 0-10 (0 no symptoms and 10 intolerable symptoms).

SECONDARY OUTCOMES:
Perceived rate of exertion | One day
  The participant will be asked to grade the exertion of 6 minutes' walk using this scale. It is a valid and reliable tool for measuring the perceived exertion in people with MS

CONTACTS AND LOCATIONS:
Overall Officials: Siva Nair, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Derived] Chotiyarnwong C, Nair K, Angelini L, Buckley E, Mazza C, Heyes D, Ramiz R, Baster K, Ismail A, Das J, Ali A, Lindert R, Sharrack B, Price S, Paling D. Effect of remote ischaemic preconditioning on walking in people with multiple sclerosis: double-blind randomised controlled trial. BMJ Neurol Open. 2020 Mar 23;2(1):e000022. doi: 10.1136/bmjno-2019-000022. eCollection 2020. PMID 33681776